CLINICAL TRIAL: NCT06609603
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-design Clinical Study to Evaluate the Body Fat Reducing Effect of Heat-Treated Green Tea Extract Complex
Brief Title: Clinical Study to Evaluate the Body Fat Reducing Effects of Heat-Treated Green Tea Extract Complex
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP-PV-2023-01
Record Dates: First submitted 2024-09-10; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Body Fat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HTGT compound (Experimental): * Dietary supplement: HTGT compound
    * oral administration of HTGT compound once daily, 2 capsules per day.
  * Dietary supplement; Placebo
    * oral administration of placebo once daily, 2 canpules per day
  Interventions: Dietary Supplement: HTGT compound
- Placebo (Placebo Comparator): Once daily, 2 capsules per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: HTGT compound — oral administration of HTGT compound once daily
  Arms: HTGT compound
Dietary Supplement: Placebo — Oral administration of placebo once daily
  Arms: Placebo

SUMMARY:
This clinical study was designed to evaluate the efficacy and safety of body fat reduction in obese adults by treatment of heat-treated green tea extract complex

DETAILED DESCRIPTION:
This study is a 12-week, randomized, double-blind, placebo-controlled clinical trial. 100 subjects were ranromly assigned to heat-treated green tea extract(HTGT) group and placebo group. The changes in the efficacy endpoint were evaluated after treatment of 2 capsules of HTGT once daiy for 12 weeks.

ELIGIBILITY:
* lt;Inclusion Criteria>

  * Males and females aged between 19 ~ 64 years
  * BMI 25.0 ~ 34.9 kg/m^2
  * Waist circumferebce: 90cm or more for men, 85cm or more for women
  * Subjects who have fully understand the information provided about the study and voluntarily decided to participate
* lt;Exclusion Criteria>

  * Participants whose weight changed by more than 10% within the 3 months prior to visit 1
  * Individuals participated in a commercial weight loss program within 3 months prior to Visit 1
  * Participants who have undergone surgical procedures within 3 years
  * Participants who have taken obesity treatment medications within the last 3 months
  * Individuals who have taken medications affecting weight or dietary supplements for weight control within the last month
  * Subjects with uncontrolled hypertension
  * Subjects diagnosed with diabetes
  * TSH <0.1 uIU/ml or >10 uIU/ml
  * Creatinine >1.5mg/dL
  * AST or ALT > three times the upper normal limit

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of body fat by DEXA | Baseline, Week 12
  Measurement was made by using dual-energy X-ray absorption(DEXA)

SECONDARY OUTCOMES:
Changes of total abdominal fat area, visceral fat area and subcutaneous fat area | Baseline, Week 12
  Measurement of the target area is made using computed tomography
Changes of indicator of lipid metabolism | Baseline, Week 12
  indicator of lipid metabolism (i.e., TC, TG, HDL, LDL)
Changes of waist circumference | Baseline, Week 12
  Measurement of waist circumfernece was performed in accordance with WHO guideline
Changes of blood biomarker | Baseline, Week 12
  adiponectin, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Wook Song, M.D./Ph.D, Principal Investigator — Catholic University St. Vincent Hospital
Locations (1):
- Catholic University St. Vincent Hospital, Suwon, Gyeonggi-do, South Korea